CLINICAL TRIAL: NCT04661514
Title: Evaluation of Psilocybin in Anorexia Nervosa: Safety and Efficacy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: COMPASS Pathways (Industry)
Responsible Party: Principal Investigator, Walter Kaye, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 049345
Record Dates: First submitted 2020-11-19; First posted 2020-12-10 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia; Anorexia Nervosa Signs and Symptoms; Eating Disorders; Mental Disorders; Psilocybin; Hallucinogens; Physiological Effects of Drugs; Psychotropic Drugs; Psychedelic Drugs
MeSH Terms: conditions — Anorexia Nervosa; Anorexia; Feeding and Eating Disorders; Mental Disorders | interventions — Psilocybin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Safety, Tolerability, and Treatment (Experimental): On dosing day, each participant will receive 1 x 25 mg treatment bottle containing 5 x 5 mg oral capsules of psilocybin. The administration session will last approximately 4-6 hours and will be supported by a lead therapist and an assisting therapist.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Psilocybin-assisted psychotherapy

SUMMARY:
The primary aim of this study is to assess the safety and tolerability of one 25 mg dose of psilocybin in participants with anorexia nervosa based on adverse events (AEs), changes in vital signs, electrocardiograms (ECGs) and clinical laboratory tests. The secondary objectives are to explore the efficacy of a single 25 mg dose of psilocybin on eating disorder symptoms and behaviors, body image, anxiety, food related obsessions and rituals, and body weight.

DETAILED DESCRIPTION:
Because there are no proven treatments that normalize core symptoms in adult anorexia nervosa, a disorder with high chronicity, many individuals seek out alternative approaches to care. Recent evidence has suggested that anxiety, obsessive compulsive disorder, and diminished reward or motivation play key roles in the development and maintenance of dysfunctional eating, and poor outcome. In recent years, a growing number of studies have demonstrated the safety and preliminary efficacy of psilocybin in clinical trials for a range of psychiatric illnesses including treatment resistant depression, obsessive compulsive disorder, addiction, and anxiety. Psilocybin may represent a promising new treatment for anorexia nervosa. However, no studies have tested psilocybin in this eating disorder population. Accordingly, this study aims to establish the safety, tolerability and dosing of psilocybin in adult patients with anorexia nervosa, as well as gather pilot data on possible efficacy.

For this study, the investigators will recruit adults who currently have a DSM-V diagnosis of anorexia nervosa. Participants will undergo medical and psychological screening and those who are deemed eligible will partake in a maximum of 7 study visits, lasting from 4-8 weeks. On dosing day, participants will receive a single 25 mg dose of psilocybin along with psychotherapeutic support, which includes preparation and integration sessions surrounding the experience. There will be a follow-up period of one month following the psilocybin session during which a range of psychological measures (questionnaires and interviews) will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 40 years of age at Screening
2. Current diagnosis of Anorexia Nervosa (informed by DSM 5) based on medical records, clinical assessment, weight, and documented completion of the version 7.0.2 Mini International Neuropsychiatric Interview (MINI)
3. Agree for the study team to maintain contact with their primary care team for the duration of the study.
4. Ability to complete all protocol required assessment tools without any assistance or alteration to the copyrighted assessments, and to comply with all study visits.

Exclusion Criteria:

Medical exclusion criteria will be determined during the Screening Period and Baseline. Exclusion assessments that will be rechecked on the day of dosing are marked with an Asterix.

1. BMI < 16 kg/m2 *
2. Medical instability as indicated by significant (>3kg) weight loss during the screening period, orthostatic heart rate and blood pressure *
3. Women who are pregnant, nursing, or planning a pregnancy in the near future. Male and female participants who are sexually active must agree to use a highly effective contraceptive method throughout their participation in the study. Women of child bearing potential must have a negative urine pregnancy test at Screening visits and Baseline, and psilocybin dosing session days *
4. Cardiovascular conditions: recent stroke (<1 year from signing of ICF), recent myocardial infarction (<1 year from signing of ICF), uncontrolled hypertension (blood pressure >140/90 mmHg) or clinically significant arrhythmia within 1 year of signing the ICF.
5. Uncontrolled or insulin-dependent diabetes.
6. Seizure disorder.
7. Use of psychedelics, including psilocybin, within one year prior to Screening assessment
8. Positive urine drug screen for illicit drugs or drugs of abuse in the Screening Period and Baseline and psilocybin dosing days. Any positive urine drug test will be reviewed with participants to determine the pattern of use and eligibility will be determined at the investigator's discretion *
9. Current enrolment in any investigational drug or device study or participation in such within 30 days prior to Screening
10. Abnormal and clinically significant results on the physical examination, vital signs, ECG, or laboratory tests at Screening, such as liver function tests (LFTs) three times greater than the upper limit of normal, reduced glomerular filtration rate (GFR) and elevated creatinin two times of upper limit of normal
11. Any other clinically significant cardiovascular, pulmonary, gastrointestinal, hepatic, renal or any other major concurrent illness that, in the opinion of the investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if he/she takes part in the study
12. Non-English speakers
13. Current or past history of schizophrenia, psychotic disorder, bipolar disorder, significant history of mania, delusional disorder, paranoid personality disorder, schizoaffective disorder, or borderline personality disorder as assessed by medical history and a structured clinical interview
14. McLean Screening Instrument for Borderline Personality Disorder >7 at Screening
15. Currently taking a serotonergic medication. All serotonergic medication must be discontinued at least two weeks prior to Baseline.
16. Current (within the last year) alcohol or substance use disorder as informed by DSM-5 at Screening
17. Significant suicide risk as defined by (1) suicidal ideation as endorsed on items 4 or 5 on the Colombia-Suicide Severity Rating Scale (C-SSRS) within the past year, at Screening or at Baseline, or; (2) suicidal behaviors within the past year, or; (3) clinical assessment of significant suicidal risk during subject interview (pre-treatment Baseline sessions).
18. Other personal circumstances and behavior judged to be incompatible with establishment of rapport or safe exposure to psilocybin, including exposure to psilocybin within the past year and use of psychedelics, such as ayahuasca, during the current episode.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Incidence and occurrence of changes in AEs | Baseline to Day 28
Incidence and occurrence of changes in AEs | Day 1 to Day 28
Incidence of clinically important changes in ECG parameters | Baseline to Day 1
Incidence of clinically important changes in ECG parameters | Baseline to Day 7
Incidence of clinically important changes in ECG parameters | Baseline to Day 28
Incidence of clinically important changes in laboratory tests | Baseline to Day 1
Incidence of clinically important changes in laboratory tests | Baseline to Day 7
Incidence of clinically important changes in laboratory tests | Baseline to Day 28
Incidence of clinically significant changes in vital signs | Baseline to Day 1
Incidence of clinically significant changes in vital signs | Baseline to Day 7
Incidence of clinically significant changes in vital signs | Baseline to Day 28
Incidence of changes in the Columbia-Suicide Severity Rating Scale (C-SSRS) at each post-Baseline visit | Baseline to Day 28
  The C-SSRS will be used to assess suicide potential or tendency as a study entry criteria and monitored throughout the study.

SECONDARY OUTCOMES:
Change in Eating Disorder Examination (EDE) scores for Dietary Restraint, Eating Concern, and Shape Concern | Baseline to Day 28
  The EDE is a structured clinical interview (investigator rated) and is used to measure the severity of the characteristic psychopathology of eating disorders. The four EDE subscales (Dietary Restraint, Eating Concern, Weight Concern, and Shape Concern) are rated on a 7-point forced-choice format (0-6), with higher scores reflecting greater severity or frequency.
Change in weight (kg) | Baseline to Day 7 and Day 28
Change in trait anxiety and state anxiety total scores on the Spielberger State-Trait Anxiety Inventory (STAI) | Baseline to Day 1, Day 7, and Day 28
  The STAI consists of self-report scales for measuring "state" and "trait" anxiety. It consists of 40 items scored by a 4 point Likert scale. 20 questions refer to state anxiety, and 20 to trait anxiety thus each section is scored between 20 and 80. Higher scores indicate greater anxiety.
Change in Physical Appearance State and Trait Anxiety Scale (PASTAS) trait total score and state score | Baseline to Day 1, Day 7, and Day 28
  The PASTAS is a self-reported 16-item measure that assesses anxiety about physical appearance. Each question is rated on a Likert scale from 0 to 4, indicating that the individual feels anxious, tense or nervous about a specific body part or general overweightness. There is a minimum score on each scale 0 and a maximum score of 64, where higher scores indicated greater severity in anxiety.
Change in Body Image State Scale (BISS) total score | Baseline to Day 28
  The BISS is a self-report questionnaire that has six items used to assess an individual's evaluative and affecting body image state at a given moment in time. The six items are: 1) dissatisfaction with physical appearance, 2) dissatisfaction with body size and shape, 3) dissatisfaction with weight, 4) feelings of physical unattractiveness, 5) current feeling about one's look relative to how one usually feels, and 6) evaluation of one's appearance relative to how the average person looks. Each item is evaluated on a 9-point bipolar Likert like scale and higher scores indicate more positive body image.
Change in Yale Brown Cornell Eating Disorder Scale (YBC-EDS-SRQ) | Baseline to Day 1, Day 7, and Day 28
  This self-report scale consists of 65 items and 19 question items related to eating disorder preoccupations and rituals. There is an emphasis on comparison between current state (last two weeks) and worst state, the one month where the participant believed their eating disorder to be the most severe. The scoring includes a preoccupations subtotal, rituals subtotal and total score.
Change in Eating Disorder Inventory (EDI) total score | Baseline to Day 1, Day 7, and Day 28
  The EDI is a self-report questionnaire. It consists of 91 items organized into 12 primary scales rated on a 0-4 point scoring system, consisting of 3 eating disorder specific scales and 9 general psychological scales that are highly relevant to, but not specific to, eating disorders. It yields six composite scores: one that is eating disorder specific (i.e., Eating Disorder Risk) and five that are general integrative psychological constructs (i.e., Ineffectiveness, Interpersonal Problems, Affective Problems, Overcontrol, General Psychological Maladjustment). A computer-based scoring program generates a detailed clinical profile and scoring report for each participant.
Change in Eating Disorder Examination Questionnaire Short Form (EDE-QS) total scores | Baseline to Day 1, Day 7, and Day 28
  The EDE-QS is a self-report questionnaire. It consists of 32 items that assess the core symptoms of eating disorders and range of eating-related psychopathology. The EDE-QS is based closely on the EDE interview. Scores range from 0 to 36 and higher scores indicate greater eating disorder symptoms.

OTHER OUTCOMES:
Change in Quick Inventory of Depressive Symptomatology (QIDS) total score | Baseline to Day 1, Day 7, and Day 28
  The QIDS is a self-reported scale. Total QIDS scores range from 0 to 27, with scores of 5 or lower indicative of no depression, scores from 6 to 10 indicating mild depression, 11 to 15 indicating moderate depression, 16 to 20 reflecting severe depression, and total scores greater than 21 indicating very severe depression.
Change in Clinical Impairment Assessment (CIA) total scores | Baseline to Day 1, Day 7, and Day 28
  The CIA is a self-reported 16-item scale of the level of social and psychological impairment that is due to eating disorder characteristics in the past 28 days. The subscales are in mood, self-perception, cognitive functioning, interpersonal functioning and work preference. The items are rated on a Likert scale with four response categories. The scores range from 0 to 48, with a higher score indicating a higher level of impairment.
Change in Visual Analogue Scales (VAS) measures | Baseline to Day 1, Day 7, and Day 28
  The VAS will be self-reported ratings of hunger, fullness and desire to eat and are designed specifically for this study. Participants will mark the degree of their experience in relation to anchors along a 100mm continuum.
Change in Eating Disorder readiness to change and motivation for change (ED-RR) | Baseline to Day 1, Day 7, and Day 28
  The ED-RR is a self-reported, two-part 18-item questionnaire that examines readiness to change in nine dimensions of eating disorder behavior (restriction, weight-shape over evaluation, binge eating, vomiting, laxative use, fasting, diuretic use, weight-gain phobia, exercise). The first part measures on a Likert scale from 1-10 the subjective readiness of the patient to change. The second part measures whether the motivation to change is for others, or the self. The scale ranges from 0% (not much for me) to 100% (mostly for me). There is also an option across both parts if the participant does not engage in a particular eating disorder behavior. Higher readiness to change has shown a correlation with a decrease in eating disorder symptoms over time.
Summary of the 5D-Altered states of consciousness questionnaire (5D-ASC) on the day of psilocybin dosing | Dosing Day
  The 5D-ASC is a self-report questionnaire. It measures the acute drug effects using five primary dimensions and respective subdimensions to assess alterations in mood, perception, and experience of self in relation to environment and thought disorder. The 5 dimensions include: oceanic boundlessness, anxious ego dissolution, visionary restructuralization, auditory alterations, and reduction of vigilance. This will be administered immediately after the psilocybin session.
Correlation between psychedelic intensity and experience and eating disorder psychopathology | Dosing Day, Day 1, Day 28
  Psychedelic intensity and experience as measured by the Five Dimension Altered States of Consciousness Questionnaire (5D-ASC); eating disorder psychopathology using the Eating Disorder Examination Questionnaire Short Form (EDE-QS)
Patient experience and acceptability of the treatment summarized | Dosing Day, Day 1, Day 28
  Summary of patient experience and acceptability of treatment will be assessed through a qualitative interview with a therapist

CONTACTS AND LOCATIONS:
Locations (1):
- Altman Clinical and Translational Research Institute, La Jolla, California, United States

REFERENCES:
- [Derived] Peck SK, Shao S, Gruen T, Yang K, Babakanian A, Trim J, Finn DM, Kaye WH. Psilocybin Therapy for Females With Anorexia Nervosa: A Phase 1, Open-Label Feasibility Study. Focus (Am Psychiatr Publ). 2024 Jul;22(3):381-387. doi: 10.1176/appi.focus.24022013. Epub 2024 Jun 28. PMID 38988455
- [Derived] Peck SK, Shao S, Gruen T, Yang K, Babakanian A, Trim J, Finn DM, Kaye WH. Psilocybin therapy for females with anorexia nervosa: a phase 1, open-label feasibility study. Nat Med. 2023 Aug;29(8):1947-1953. doi: 10.1038/s41591-023-02455-9. Epub 2023 Jul 24. PMID 37488291